CLINICAL TRIAL: NCT06635057
Title: A Phase 4, Multicenter, Multi-Country, Open-Label, Single-Arm Study to Investigate the Effectiveness and Safety of Tirzepatide Once Weekly in Adult Participants With Type 2 Diabetes During Ramadan
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Type 2 Diabetes During Ramadan
Acronym: T-RAM
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27195; I8F-MC-GPIY (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-10-04; First posted 2024-10-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Ramadan; Fasting
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fasting | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tirzepatide (Experimental): Participants will receive tirzepatide subcutaneously (SC)
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176

SUMMARY:
The main purpose of the study is to investigate whether tirzepatide can be effectively started before Ramadan and used per label in participants with Type 2 Diabetes during the fasting month.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of uncontrolled Type 2 Diabetes based on the World Health Organization classification or other locally applicable diagnostic standards, and who intend to fast during Ramadan
* Have HbA1c ≥7% within 30 days prior to screening
* Are glucagon-like peptide-1 receptor agonist (GLP-1 RA) naïve
* Have had stable body weight self-reported change ≤5 kilograms (kg) during the 90 days prior to screening
* Have body mass index ≥25 kilograms per square meter (kg/m2) at screening

Exclusion Criteria:

* Have Type 1 Diabetes or gestational diabetes
* Have a history of chronic or acute pancreatitis
* Have acute or chronic hepatitis
* Have evidence of a significant, uncontrolled endocrine abnormality
* Have a history of an active or untreated malignancy
* Have New York Heart Association Functional Classification IV congestive heart failure
* Have been treated with insulin within two weeks prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline (20 to 8 weeks Before Ramadan), Week 4-8 from Start of Ramadan (SoR)

SECONDARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline (20 to 8 weeks Before Ramadan), Week 4-8 from SoR
Number of Hypoglycemic Events | Baseline (20 to 8 weeks Before Ramadan), Week 4-8 from SoR
Number of Self-Reported Gastrointestinal (GI) Adverse Events | Baseline (20 to 8 weeks Before Ramadan), Week 4-8 from SoR
Percentage of Participants Achieving HbA1c <7% | Baseline (20 to 8 weeks Before Ramadan), Week 4-8 from SoR
Change from SoR to End of Ramadan (EoR) in the 5-Level European Quality of Life 5 Dimensions (EQ-5D-5L) | SoR (Week 0), EoR (Week 4)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- Saudi Arabia (15):
  - Al Moosa Specialist Hospital, Al Ahasa
  - National Guard Hospital-King Abdulaziz Medical City, Alahsa
  - King Abdulaziz Medical City-Jeddah, Jeddah
  - King Fahad Armed Forces Hospital Jeddah, Jeddah
  - King Faisal Specialist Hospital & Research Center, Jeddah
  - Saudi Airlines Medical services, Jeddah
  - King Faisal Specialist Hospital and Research Center Madina, Madinah
  - King Saud University, Riyadh
  - Osepdale Fatebenefratelli e Oftalmico, Riyadh
  - Al Dallah Hospital, Riyadh
  - Sulaiman Habib Olaya, Riyadh
  - Specialized Medical Center Hospital, Riyadh
  - Dallah Namar Hospital, Riyadh
  - Dr. Sulaiman Al Habib Hospital As Suwaidi, Riyadh
  - Dr. Sulaiman Al Habib Medical Complex Arrayan Saudi Arabia, Riyadh
- United Arab Emirates (14):
  - Lifecare Hospital, Abu Dhabi
  - Tawam Hospital, Abu Dhabi
  - Imperial College London Diabetes Center, Abu Dhabi
  - NMC Abu Dhabi, Abu Dhabi
  - Rashid Centre for Diabetes and Research, Ajman
  - Thumbay University Hospital, Ajman
  - Emirates Hospital Dubai, Dubai
  - Aster Clinics, Dubai
  - Dubai Diabetes Center, Dubai
  - Dubai Hospital, Dubai
  - Medcare Hospital, Dubai
  - Mediclinic City Hospital, Dubai
  - Rashid Hospital., Dubai
  - Medcare Hospital, Sharjah city

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/